CLINICAL TRIAL: NCT06374615
Title: Insights Into Tick-Borne Diseases: a Prospective Study From an Endemic Area of Northern Italy
Brief Title: Insights Into Tick-Borne Diseases: a Study From an Endemic Area of Northern Italy
Acronym: TICKTOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-07
Record Dates: First submitted 2024-04-11; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Tick-Borne Diseases
MeSH Terms: conditions — Tick-Borne Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serological test for Tick-borne Patogens (Experimental): A baseline visit (T0) will be scheduled within 7-10 days of the tick bite. T0 visit will include: signature of ICF, data collection, blood sampling. Signature of a specific consent will be sought for storage of the leftover samples at -80°.
  12 weeks apart from the bite (T1), subjects will be invited to a clinical and serological follow-up visit.
  Participants will be taught to contact the study investigators in case of emergence of compatible signs/symptoms. In this case, one of the study members will call the participant to schedule an additional visit (T unscheduled, TU). At this time a blood sample will be collected. Timing for molecular and serological tests will be performed in relation to the emergence of patient's symptoms. In case of TBDs caused by TBEV, Rickettsia spp, Borrelia spp, Ehrlichia, Anaplasma spp. and Babesia spp the patient will be treated according to standard clinical practice.
  Interventions: Diagnostic Test: IgG and IgM search for specific Tick-Borne Patogens

INTERVENTIONS:
Diagnostic Test: IgG and IgM search for specific Tick-Borne Patogens — Ticks will be classified based on morphological characteristics by microscopy observation.
  For TBP detection by molecular test, Nucleic acid extraction will be performed on ticks lysate or blood using kits MagMAX TM Viral/Pathogen Nucleic Acid Isolation Kit (Thermo Fisher Scientific) on MagEX STARlet platform from Hamilton. Species identification by molecular method will be performed by Sanger sequencing for Rickettsiae and Babesia, and Multi-Locus Sequence Typing will be used to characterize Borrelia.
  Serum samples collected throughout the study will be tested to assess any seroconversions during the follow-up period.
  Samples will be tested for the presence of specific IgG and IgM for the following TBPs: TBEV, R. typhi. R. conorii, Borrelia spp, Anaplasma, Ehrlichia and Babesia.

SUMMARY:
This is a monocentric, experimental, non-pharmacological and non-device no profit study.

The study is experimental because all the visits and blood withdrawals foreseen by the protocol do not fall within the normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* all individuals aged > 8 years presenting for tick removal.
* Individuals providing signed informed consent.

Exclusion Criteria:

* tick not available for analysis

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of individuals diagnosed with Tick-Borne Diseases (TBD) over the total number of individuals who were bitten by a tick which carried an identified TBP. | baseline

SECONDARY OUTCOMES:
Number of identified Tick-Borne Patogenees (TBPs) on the total number of analyzed ticks | baseline
Number of individuals who developed symptoms and were diagnosed for a TBP infection during the 12 weeks' follow-up period | 12 weeks
Number of individuals who developed specific antibodies against a TBP after tick bite. | 12 weeks
List of novel TBPs that were not previously found in the study areas. | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Sacro Cuore Don Calabria hospital, Negrar, Verona, Italy